CLINICAL TRIAL: NCT05242679
Title: Effect of Myofascial Release With Tennis Ball on Spasticity and Upper Limb Motor Functions in Patients With Chronic Stroke
Brief Title: Effect of Myofascial Release With Tennis Ball on Spasticity and Motor Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GSTIESC/23/16
Record Dates: First submitted 2022-02-06; First posted 2022-02-16 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Stroke
Keywords: Myofascial release; Chronic stroke; Motor functions; Spasticity; modified Ashworth scale; Fugl-Meyer assessment scale
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: Two-arm parallel pre-test-post-test experimental design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release Group (Experimental): Participants were treated with a conventional physiotherapy program along with myofascial release with a tennis ball.
  Interventions: Other: Myofascial release technique along with conventional physiotherapy exercises
- Conventional Physiotherapy Group (Active Comparator): A conventional physiotherapy program was provided including range of motion/flexibility exercises, strength training, postural control, functional mobility exercises, lower limb functional exercises, and gait training.
  Interventions: Other: Conventional physiotherapy exercises

INTERVENTIONS:
Other: Myofascial release technique along with conventional physiotherapy exercises — Myofascial release technique was performed using a tennis ball along with conventional physiotherapy exercises.
  Arms: Myofascial Release Group
Other: Conventional physiotherapy exercises — Conventional physiotherapy exercises were performed including the range of motion/flexibility exercises, strength training, postural control, functional exercises, and gait training.
  Arms: Conventional Physiotherapy Group

SUMMARY:
Impaired motor function and upper extremity spasticity are common concerns in patients after stroke. It is essential to plan therapeutic techniques to recover from the stroke. The objective of this study was to investigate the effects of myofascial release with the tennis ball on spasticity and motor functions of the upper extremity in patients with chronic stroke.

DETAILED DESCRIPTION:
Myofascial release is a therapeutic technique that aims to improve flexibility and sliding between layers of soft tissues, reduce the severity of muscle activity pain, and improve functional performance. A previous study included myofascial release with a tennis ball in the lower extremity in patients with chronic stroke and reported improved balance. Different other unique therapeutic interventions have been proposed over the past two decades for stroke management; however, myofascial release with a tennis ball has not been included in them. Therefore, the present study aimed to examine the effects of myofascial release with a tennis ball on spasticity and motor functions of the upper limb in patients with chronic stroke.

Participants were equally divided into two groups viz. experimental and control, with 11 participants in each group.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke,
* Hemiplegia with upper extremity dysfunctions of more than 6 months and less than 2 years of duration
* modified Ashworth scale of grade 1-3,
* Mini-Mental State Exam (MMSE) >24 suggesting intact cognition,
* full passive range of motion of the shoulder, elbow, wrist, and hand joints
* voluntary control by Brunnstrom of grade 3-5 for shoulder, elbow, and wrist joints

Exclusion Criteria:

* circulatory problems such as deep vein thrombosis,
* impaired sensation over the affected upper limb,
* recently injured area/open wounds,
* arthritic or any other musculoskeletal condition of the upper extremity, shoulder instability based on the posterior or anterior apprehension test, and positive sulcus test,
* history of brain surgery after stroke,
* Botox injection in the past four months,
* medically unstable patients,
* patients who have had multiple strokes.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2017-10-23 (Actual)

PRIMARY OUTCOMES:
Spasticity | 4 weeks.
  Spasticity measured using Modified Ashworth scale - Scores range from 0 to 4, where lower scores represent normal muscle tone and higher scores represent spasticity.
Upper limb motor functions | 4 weeks.
  Upper limb motor functions measured using Fugl-Meyer Assessment Scale - Scores range from 0-66, where lower score represent poor performance of upper extremity and higher scores represents good performance of upper extremity

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parikh RJ, Sutaria JM, Ahsan M, Nuhmani S, Alghadir AH, Khan M. Effects of myofascial release with tennis ball on spasticity and motor functions of upper limb in patients with chronic stroke: A randomized controlled trial. Medicine (Baltimore). 2022 Aug 5;101(31):e29926. doi: 10.1097/MD.0000000000029926. PMID 35945719